CLINICAL TRIAL: NCT07105488
Title: A Phase 2, Parallel-arm, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study to Evaluate the Efficacy and Safety of BFB759 in Patients With Atopic Dermatitis (COMPASS 2-AD)
Brief Title: A Study Evaluating BFB759 in Moderate to Severe Atopic Dermatitis
Acronym: COMPASS 2-AD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Bluefin Biomedicine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL-BFB759-002
Record Dates: First submitted 2025-07-21; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis (AD)
Keywords: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Intervention Model Description: Parallel-arm, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Active - high dose (Experimental): BFB759 high dose Day 1 followed by BFB759 every 2 weeks (Q2W) starting at Week 2 through Week 14 (inclusive), which is followed by placebo Q2W at Weeks 16 through 30 (inclusive)
  Interventions: Biological: BFB759
- Placebo (Placebo Comparator): Placebo Q2W for 14 weeks. At Week 16, participants in Placebo group who are still enrolled in the study and receiving treatment will be re-randomized (1:1) into two groups (Cross-1 or Cross-2) to receive BFB759 intervention.
  * Cross-1 will receive BFB759 at Week 16, and then BFB759 Q2W at Week 18 through Week 30 (inclusive).
  * Cross-2 will receive BFB759 at Week 16, and then BFB759 Q2W at Week 18 through Week 30 (inclusive).
  Interventions: Biological: BFB759; Drug: Placebo
- Active - low dose (Experimental): BFB759 low dose on Day 1 followed by BFB759 every 2 weeks (Q2W) starting at Week 2 through Week 14 (inclusive), which is followed by placebo Q2W at Weeks 16 through 30 (inclusive)
  Interventions: Biological: BFB759

INTERVENTIONS:
Biological: BFB759 — BFB759 is a human mAb that inhibits multiple pro-inflammatory cytokines that contribute to the pathogenesis of multiple disease processes characterized by aberrant inflammation, including atopic dermatitis
Drug: Placebo — Placebo for BFB759
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled study where subjects are participating for approximately 36 to 40 weeks. The study compares how well BFB759 works and how safe it is compared with a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Are adults (18-75) with a diagnosis of atopic dermatitis for at least one year.
* Have moderate to severe disease not adequately controlled by topical treatments.
* Are willing to follow study instructions, attend regular visits, and avoid certain other medications during the study.

Exclusion Criteria:

* Have certain infections or other immune conditions.
* Recently used medications that could interfere with the study.
* Are pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of BFB759 in AD | week 16 and week 32
  To evaluate the efficacy of BFB759 in adult male and female participants with AD as assessed by Eczema Area and Severity Index (EASI) score. Measure improvements in redness, swelling, scratching damage, and roughness.

SECONDARY OUTCOMES:
How well the treatment works at Week 16 | Week 16
  * How many participants had at least a 50%, 75%, or 90% improvement in their eczema signs.
  * How much the severity and size of eczema-affected areas improved.
  * Whether participants felt less itchy.
  * How many participants had a drop of 4 or more points in their itch score (especially for those who started with a higher itch level).
How well the treatment works at week 32 | Week 32
  * How much eczema signs changed from Week 16.
  * How many participants had a 50%, 75%, or 90% improvement since Week 16.
  * Changes in eczema severity and itch compared to Week 16.
  * How many people had a 4-point drop in their itch score (again, only among those who had higher itch scores at Week 16).
Safety and tolerability | 21 months (about 22 visits during the course of study)
  * record side effects and severity
  * record how well participants tolerate the treatment over time

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Antelope Valley Clinical Trials, Lancaster, California
  - Ziaderm Research LLC, North Miami Beach, Florida
  - Conquest Research LLC, Winter Park, Florida
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Vitality Clinical Trials LLC, Woodbury, New York
  - Apex Clinical Research Center, LLC, Mayfield Heights, Ohio
  - Stryde Research-Epiphany Dermatology, Southlake, Texas

IPD SHARING:
Plan to Share IPD: No